CLINICAL TRIAL: NCT06035458
Title: Potential Osteocatabolic Effect Caused by Anti-CGRP mAbs in Migraine Patients Treated With Anti-CGRP mAbs - an Observational Pilot Project With Prospectively Collected Health Related Data
Status: Active, not recruiting | Type: Observational
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Chiara Zecca, Prof, Ente Ospedaliero Cantonale, Bellinzona
Other Study IDs: EOCNSIHA_2201
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Migraine Disorders
Keywords: Migraine; anti-CGRP mAb; Densitometry; osteocatabolic effect
MeSH Terms: conditions — Migraine Disorders | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Diagnostic radiology — Clinical procedures include bone mineral measurement (bone densitometry, dxa) performed according to clinical practice; venipunctures for laboratory assessments (haematology and blood chemistry; bone turnover biomarkers P1NP and CTX).

SUMMARY:
Background: To gain insight on the osteoanabolic activity of anti-CGRP mAbs in patients with migraine as this was not yet specifically investigated in registration or post-approval clinical studies, however, being pathophysiologically plausible. If a clinically relevant, osteocatabolic effect caused by anti-CGRP mAbs will be demonstrated by the present investigation monitoring and mitigating strategies might be required and addressed in dedicated future studies. Objectives: To investigate whether treatment with anti-CGRP mAbs over 6, 12, and 24 months is associated with changes in bone density, structure and/or metabolic turnover in migraine patients.

Project Design and Procedures: Prospective collection of health-related clinical data, open label, controlled pilot study. Demographic (ethnicity, age, sex) and physical (age, height) data, data on medical and migraine history will be collected. Clinical procedures include bone mineral measurement (bone densitometry, dxa) performed according to clinical practice; venipunctures for laboratory assessments (haematology and blood chemistry; bone turnover biomarkers P1NP and CTX).

DETAILED DESCRIPTION:
Migraine is a chronic and often lifelong disease defined by recurrent unprovoked headache episodes lasting over four hours with one or more disabling symptoms including nausea, vomiting, dizziness, and extreme sensitivity to sound and light. It directly affects more than 1 billion people worldwide, representing the most common neurological condition with an estimated 1-year prevalence of 15%. It is approximately twice as high in females compared to males. In individuals younger than 50 years, migraine represents the leading cause of years lived with disability worldwide, and a major public health concern, as it is insufficiently recognized leading to considerable individual and societal costs. The current migraine treatment armamentarium available includes acute and preventive medications, as well as non-pharmacological approaches. Preventive therapies used until recently were just non-specific medications such as beta-blockers, calcium channel antagonists, antidepressants, and antiepileptic drugs, which are often limited by insufficient efficacy and/or relevant short and long-term side effects. More recently, anti-calcitonin gene related peptide (CGRP) monoclonal antibodies (mAbs) have been approved as pharmacological preventive therapies for migraine and currently represent game changer in the field. CGRP, a 37-residue neuropeptide produced in specific neurons by alternative splicing of the calcitonin gene, acts as a potent vasodilator as well as a neurotransmitter. In humans, CGRP is present in two isoforms, α-CGRP and β-CGRP. α-CGRP is the principal isoform localized in the peripheral and central sensory nervous system, and plays a key role in the underlying mechanism of migraine, as illustrated by several lines of preclinical and human evidence. Intravenous infusion of this neuropeptide elicits vasodilatation and precipitates migraine attacks in subjects diagnosed with migraine. Additionally, an increase in plasma CGRP concentrations can be measured in the craniovascular circulation during migraine attacks. At the trigeminocervical complex, CGRP also plays a crucial role in central sensitization, a critical step in the development of migraine headache. Accordingly, blockade of the CGRPergic transmission has become attractive for the development of targeted and highly effective migraine treatment strategies. These include mAbs binding CGRP (galcanezumab, fremanezumab, eptinezumab), or its receptor (CGRPR; erenumab). When used as preventive therapies in patients with episodic or chronic migraine, these new antimigraine mAbs (anti-CGRP mAbs) showed effectiveness in reducing the frequency and intensity of attacks and as well as migraine associated symptoms. Anti- CGRP mAbs were well-tolerated and safe according to pivotal trials and their open label extensions up to 5 years. The most frequent adverse events reported in these studies were nasopharyngitis, upper respiratory tract infections, nausea, arthralgia, fatigue, and injection site pain, however these did not generally exceed rates observed in placebo treatment arms. However, patients included in registration clinical trials may differ from those treated in the clinical practice, since the former are typically limited in number, younger, and with a low burden of comorbidities and concomitant medications. Consequently, the adverse event profile of a given drug can significantly differ in these two contexts, underlining the importance of post-marketing surveillance and 'real world' observational studies. According to that, in clinical trials the administration of anti-CGRP mAbs did not produce significant cardiovascular side effects, which represented a concern since CGRP is a potent physiological vasodilator widely represented in the human body. Instead, the first-inclass mAb erenumab was recently found to be associated with an increased risk of new onset or worsening arterial hypertension, which has now been included among warnings in the the erenumab label by FDA. Based on the wide distribution of CGRP and its receptor in the body, additional off-target effects might be also expected when anti-CGRP mAbs are used extensively in the clinical practice. Besides the cardiovascular system, the CGRP/CGRP receptor system is actually present in the central and peripheral nervous system (particularly, the blood brain barrier, the anterior pituitary, the pineal gland, and the area postrema), gastrointestinal and vestibular system, the kidney and the skin, and has a role in the endocrinal system and bone metabolism.

The objective of this study is to investigate whether treatment with anti-CGRP mAbs over 6, 12, and 24 months is associated with changes in bone density, structure and/or metabolic turnover in migraine patients.

We hypothesize that the continuous use of anti-CGRP mAbs causes bone reabsorption, which in turn reflects in increased bone catabolic biomarkers, decreased bone anabolic biomarkers and ultimately in reduced bone density (BMD) and altered trabecular structure (TMS).

ELIGIBILITY:
Inclusion Criteria:

Anti-CGRP mAbs treated group (TC):

* Anti-CGRP mAbs naïve males and females;
* Aged between 18 and 50 years;
* Affected with migraine with or without aura [4];
* Planning to start a migraine preventive monotherapy with and satisfying the prescription criteria for Anti-CGRP mAbs erenumab, galcanezumab, and fremanezumab according to the Swiss reimbursement authorities (previous treatment with at least 2 migraine preventive therapies among beta-blockers, calcium antagonists, anticonvulsants and selective serotonin reuptake inhibitors SSRI must have been ineffective, contraindicated or not tolerated; mean number of monthly migraine days (MMD) in three consecutive months must be at least 8).

Control group, not treated with anti-CGRP mAbs (CG)

* Males and females
* Aged between 18 and 50 years;
* Affected with migraine with or without aura [4];
* Under no migraine preventive therapies;
* Never treated with / not planning to start on anti-CGRP mAbs

Exclusion Criteria:

* An ongoing treatment with one of the following drugs: protonic pump inhibitors, selective serotonin reuptake inhibitors (such as escitalopram, fluoxetine, paroxetine, sertraline), glitazones, anti-aromatase, anti-androgen medications, glucocorticoids; having ever received glucocorticoids at doses of ≥5 mg (or equivalent) for ≥3 months, anti-retroviral drugs, vitamin k inhibitors or bone antiresorptive therapy;

  * An ongoing supplementation with calcium, vitamin D;
  * Being affected with osteoporosis or previous unprovoked fractures at adult age;
  * Being affected with significant comorbidities potentially interfering with bone metabolism including: type 1 or 2 diabetes; gastrointestinal malabsorption and/or chronic inflammatory bowel diseases; primary hyperparathyroidism; hyperthyroidism; prolonged immobilization; rheumatoid arthritis; chronic obstructive bronchopneumopathy; Cushing syndrome; any other relevant diseases according to the investigator's judgement;
  * A history of drug or alcohol abuse, or illicit substances use;
  * Hypogonadism;
  * Menopause;
  * Pregnancy or breastfeeding.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Patients who present with migraine at the Headache out-patient clinic, Neurocenter of Southern Switzerland, EOC, will be recruited during routine clinical evaluations. At our Headache Clinic, migraine patients planned to start an anti-CGRP mAb undergo a preliminary screening to identify those suffering from or at increased risk of osteoporosis/osteopenia.
  Patients not planned to start an anti-CGRP mAb will be screened to match a treated patient for age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in bone mineral density | 6-12 months
  Change in lumbar spine, total hip and femoral neck bone mineral density and lumbar spine TBS during anti-CGRP mAb.

CONTACTS AND LOCATIONS:
Locations (1):
- Chiara ZECCA, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No